CLINICAL TRIAL: NCT06877559
Title: Analysis of the Safety and Efficacy of Balloon-Assisted Enteroscopic Treatment for Phytobezoar
Brief Title: Balloon-Assisted Enteroscopic Treatment for Phytobezoar
Status: Active, not recruiting | Type: Observational
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Xiuli Zuo, Director of gastroenterology department, Shandong University
Other Study IDs: 2025-SDU-Qilu-02
Record Dates: First submitted 2025-03-10; First posted 2025-03-14 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Phytobezoar; Intestine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients who underwent balloon-assisted enteroscopic treatment for phytobezoar: Patient information was retrieved and collected through the HIS (Hospital Information System) and endoscopy system of Qilu Hospital of Shandong University, followed by statistical analysis. The collected information includes: gender, age, comorbid conditions, symptoms, time of onset, laboratory test results, time of small intestinal endoscopy, description of endoscopic procedures, success of the procedure, whether sodium bicarbonate was injected, presence of complications during treatment, length of hospital stay, and days from surgery to discharge.
  Interventions: Other: balloon-assisted enteroscopic treatment for phytobezoar

INTERVENTIONS:
Other: balloon-assisted enteroscopic treatment for phytobezoar — The endoscopists applied balloon-assisted enteroscopy for the treatment of the phytobezoar

SUMMARY:
By reviewing a case series of patients who underwent balloon-assisted enteroscopic treatment for phytobezoar at our hospital, we analyzed the safety and efficacy of this technique.

ELIGIBILITY:
Inclusion Criteria:

* Retrospectively collect data from patients who underwent balloon-assisted enteroscopic treatment for phytobezoar at our hospital.

Exclusion Criteria:

* Patients with incomplete clinical data.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: patients with small intestinal phytobezoar
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of Balloon-Assisted Enteroscopic treatment for Phytobezoar | 3 months
  Success Rate of the Procedure

SECONDARY OUTCOMES:
Safety of Balloon-Assisted Enteroscopic treatment for Phytobezoar | 3 months
  Incidence of Complications

CONTACTS AND LOCATIONS:
Overall Officials: Xiuli Zuo, Study Director — Qilu Hospital of Shandong University
Locations (1):
- Qilu hospital of shandong university, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No